CLINICAL TRIAL: NCT01324687
Title: Study Of Telemedicine Consultation at Home For Older Adults
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manish Shah, Associate Professor, University of Rochester
Other Study IDs: 31563; R01HS018047 (AHRQ)
Record Dates: First submitted 2010-11-19; First posted 2011-03-29 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-04

CONDITIONS: Physical Disorders; Telemedicine
Keywords: Telemedicine; Geriatrics
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Group without access to telemedicine in the home for acute care issues.
- Telemedicine care: Cohort with access to telemedicine in the home for acute care issues.
  Interventions: Other: Telemedicine care

INTERVENTIONS:
Other: Telemedicine care — Availability of telemedicine
  Other Names: Telemedicine
  Groups: Telemedicine care

SUMMARY:
The system of medical care for older adults with acute illnesses often serves them poorly. Many factors limit these patients' access to safe, patient-centered, efficient, high-quality, acute care. These factors include a shortage of geriatricians and primary care physicians; limited availability of timely, acute-illness, patient appointments; emergency department (ED) crowding; interruptions to the continuity of care when patients use the ED; and poor transitions of care from the ambulatory setting to the ED. These conditions foster unnecessary ED use, adverse events in the ED for which older adults are particularly at-risk, and unnecessary medical costs. As the population ages, the magnitude of these problems will only increase.

The overarching study goals are to develop and evaluate a telemedicine-enhanced care model that improves access to safe, high-quality, acute illness care for older adults; fosters appropriate use of health services; and reduces unnecessary expenditures. Specifically, this study aims to:

1. Expand the existing pediatric HeA telemedicine network to older adults by providing senior living communities (SLC) with an alternative on-site care option for individuals with an acute illness episode.

   Hypothesis 1: 90% of requested telemedicine visits will be successfully completed.
2. Evaluate the impact of the HeA telemedicine model on utilization, quality of care, and patient safety.

   Hypothesis 2: The rate of ED use will be lower at SLCs with access to care via telemedicine, as compared to SLCs without such access to care.

   Hypothesis 3: Quality of care and patient safety measures will be better for SLC residents with access to telemedicine-enhanced care than for residents without this form of access.
3. Evaluate the economic benefit of the care delivered through the telemedicine network.

   Hypothesis 4: The net cost of healthcare per patient-month will be less for SLC residents with access to telemedicine-enhanced care than for those without this form of access.
4. Use qualitative methods to identify strategies and assets that promote and conditions that impede the implementation, acceptance, and success of the HeA telemedicine network in SLCs. This knowledge will inform efforts to develop a toolkit to be used to disseminate this technology broadly.

DETAILED DESCRIPTION:
Telemedicine is a potential solution with demonstrated effectiveness in other vulnerable populations. Previous work by members of this research team has shown that telemedicine is an effective health information technology solution to address similar challenges in multiple vulnerable populations, demonstrating both improved access to care and reduced ED visits. The existing telemedicine program in Rochester, Health-e-Access (HeA), has been both successful and sustained, and well accepted by all key stakeholders including patients, families, clinicians, and insurers. This existing program, combined with the experience and multidisciplinary expertise of the investigators research team, creates a unique opportunity to (1) develop a model of care that leverages this technology to improve geriatric acute care, (2) evaluate this model through a prospective cohort study, and (3) identify key barriers and drivers of implementation to promote dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Strong Health Geriatrics Group practice
* Consent to participate
* Resident of facility with telemedicine established

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults residing in senior living communities.
Sampling Method: Non-Probability Sample
Enrollment: 1537 (Actual)
Dates: Start 2010-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish N. Shah, MD, Principal Investigator — University of Rochester; Kenneth McConnochie, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We excluded 15 individuals from analysis because they left the facility and the study less than 1 month after starting, and they were significantly different than the rest of the population. We felt that they has been mistakenly accepted into an independent or assisted living and recognized this and moved out to an alternate level of care.
Period: Overall Study
Arm/Group | Control | Telemedicine Care
Started | 1058 | 494
Completed | 1058 | 479
Not Completed | 0 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Telemedicine Care | Total
Number analyzed (Participants) | 1058 | 479 | 1537
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 85 [79 to 90] | 85 [19 to 89] | 85 [79 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 746 | 347 | 1093
  Male | 312 | 132 | 444
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 27 | 63
  White | 1022 | 452 | 1474
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1058 | 479 | 1537

OUTCOME MEASURES:

1. Primary Outcome: Emergency Department Use
Description: Use of emergency department by individuals with access to care via telemedicine as compared to those without such access to care.
Time Frame: Up to 42 months
Measure: Number; unit: Emergency dept use rate per person-month
Arm/Group | Control | Telemedicine Care
Number analyzed (Participants) | 1058 | 479
Emergency dept use rate per person-month | 0.1050 | 0.0885
Statistical Analysis 1: Comparison: Control vs Telemedicine Care; Rate ratio of ED use rate of the intervention group as compared to the control group; Test type: Superiority or Other; p = 0.017, GEE / Poisson regression models; Rate ratio = 0.8387, 95% CI 2-sided [0.7261 to 0.9689]

2. Secondary Outcome: Cost of Care
Description: Comparison of cost of care between intervention and control groups.
Time Frame: Up to 36 months
Population: The cost data was not available from the Finance Office from Rochester General Hospital or Thompson Hospital so this analysis was not performed.
Arm/Group | Control | Telemedicine Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control | Telemedicine Care
Serious Adverse Events (participants affected / at risk) | 0/1058 | 0/479
Other Adverse Events (participants affected / at risk) | 0/1058 | 0/479

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No